CLINICAL TRIAL: NCT02480595
Title: ARCHYTAS: AAA Registry: Clinical Outcomes of Highly Angulated anatomY Treated With the Aorfix™ Stent Graft
Brief Title: AAA Registry: Clinical Outcomes of Highly Angulated anatomY Treated With the Aorfix™ Stent Graft
Acronym: ARCHYTAS
Status: Suspended | Type: Observational
Why Stopped: Recruitment on hold
Sponsor: Lombard Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: ARCHYTAS
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal Aortic Aneurysm; AAA; Endovascular; EVAR; Stent; Stent Graft; High Angle; Tortuous
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EVAR: Patients undergoing endovascular repair with the latest generation Aorfix™ AAA Flexible Stent Graft System for treatment of abdominal aortic and aorto-iliac aneurysms where the aorta in the aneurysm neck is bent through an angle between 0° and 90°
  Interventions: Device: Stent Graft

INTERVENTIONS:
Device: Stent Graft — Endovascular repair of abdominal aortic aneurysm (EVAR)
  Other Names: Aorfix™ stent; Aorfix™ stent graft

SUMMARY:
The ARCHYTAS Registry is a long-term, global, multicenter, non-randomized, prospective, registry designed to collect "on-label" data in real world clinical settings on patients undergoing endovascular repair with the latest generation Aorfix™ AAA Flexible Stent Graft System. Registry data will augment existing data from ongoing and prospective Aorfix™ clinical trials for the purposes of publication, general product development and quality measures.

DETAILED DESCRIPTION:
The ARCHYTAS Registry is a long-term, global, multicenter, non-randomized, prospective, registry established by Lombard Medical Ltd. (Lombard) to collect "on-label" data in real world clinical settings on patients undergoing endovascular repair with the latest generation Aorfix™ AAA Flexible Stent Graft System, for treatment of abdominal aortic and aorto-iliac aneurysms in anatomy where the aorta in the aneurysm neck is bent through an angle between 0° and 90°. This indication for Aorfix™ is approved in all territories where this Registry is being operated and this Registry does not seek to collect data on any use of the implant for which full commercial approval does not already exist.

The ARCHYTAS Registry data will augment existing data from ongoing and prospective clinical trials with Aorfix™ for the purposes of publication, general product development and quality measures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed abdominal aortic aneurysm with indication for endovascular repair.
2. Intention to electively implant the Aorfix™ Stent Graft System.

Exclusion Criteria:

1. Does not comply with the indications for Aorfix™ in the Instructions for Use (IFU).
2. Unwillingness or inability to comply with the recommended follow-up assessments according to the standards of care at the investigative site.
3. Unwillingness or inability to provide informed consent to both the Registry and the EVAR procedure.
4. Patients in whom Aorfix™ is being placed as a secondary procedure to a previous surgical or endovascular treatment of an AAA other than with another Aorfix™ graft.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The ARCHYTAS Registry will meet objectives only if appropriate patients are enrolled. Patients presenting with AAA who fulfill inclusion criteria and are not ruled out by exclusion criteria will be included. Each investigator will record all potential participants screened for inclusion and document reasons for ineligibility. The implanting physician will consider all relevant medical and nonmedical factors when determining if a particular patient is suitable for inclusion in the Registry. In order to prevent selection bias, sites will be asked to screen and enroll patients consecutively. In circumstances where patients are screened and subsequently enrolled, but for various reasons are not implanted with the Aorfix™ device, only the screening and procedural data will be collected.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-04; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | 12 months
  Defined as freedom from the following:
  * Sac expansion > 5mm
  * Type I and III endoleaks requiring re-intervention
  * Rupture
  * Conversion to open surgery
  * Stent graft migration > 10 mm
  * Stent graft occlusion

SECONDARY OUTCOMES:
Graft Performance | 30 Days to 12 Months
  Defined as:
  * Stent graft migration > 10mm (12 months)
  * Stent graft patency (12 months)
  * Stent graft endoleaks (30 days and 12 months)
  * Aneurysm-related secondary procedure (12 months)
  * Adverse device effects (12 months)
  * Technical observations (12 months)
  * Aneurysm-related mortality (12 Months)
  * All-cause mortality (30 days and 12 months)
  * Major Adverse Events (MAEs) (30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Riambau, Principal Investigator — University Clinic, Barcelona, Spain
Locations (37):
- Prague University Hospital, Prague, Czechia
- Germany (12):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Herzzentrum Köln, Cologne
  - Alfried Krupp Krankenhaus, Essen
  - Elisabeth-Krankenhaus Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Hospital Halle, Halle
  - Universitätsklinikum Leipzig, Leipzig
  - St.Vincenz-Krankenhaus Limburg, Limburg
  - Bonifatius Hospital, Lingen
  - Klinikum Rechts der Isar der TU München, München
  - Ammerland Klinik GmbH, Westerstede
  - Universitätsklinikum Würzburg, Würzburg
- Italy (6):
  - Ospedale Papa Giovanni 23, Bergamo
  - Sant'Anna, Como
  - Ospeale Maggiore, Lodi
  - Ospedale Sant'Andrea delle Fratte, Perugia
  - Tor Vergata, Rome
  - Policlinico San Donato IRCCS, San Donato
- Auckland Hospital, Auckland, New Zealand
- Spain (9):
  - University Clinic, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - H. Universitari Dr. Josep Trueta, Girona
  - University Hospital S. Cecilio, Granada
  - HGU Gregorio Marañon, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - H. Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Donostia, San Sebastián
  - H. Marqués de Valdecilla, Santander
- United Kingdom (8):
  - Royal Bournemouth General Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - Mid Essex Hospital - Broomfield, Chelmsford
  - Northwick Park Hospital, Harrow
  - Kings College Hospital NHS Foundation Trust, London
  - Norfolk & Norwich University Hospital, Norwich
  - Nottingham University Hospital, Nottingham
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lombard Medical Home Page — http://www.lombardmedical.com